CLINICAL TRIAL: NCT02137577
Title: Prospective, Multi-center and Randomized Controlled Clinical Study to Verify Effectiveness and Safety of Drug-eluting Balloon in PTA Procedure of the Infrapopliteal Artery
Brief Title: AcoArt Ⅱ/ BTK China: Drug-eluting Balloon for Below-The-Knee Angioplasty Evaluation in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: acotec-03
Record Dates: First submitted 2014-05-05; First posted 2014-05-14 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Artery Disease
Keywords: drug eluting balloon catheter
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEB catheter (Experimental): use DEB catheter(trade name: Lotus/Tulip) to treat the stenosis or occlusion in below popliteal artery of experimental arm
  Interventions: Procedure: DEB catheter
- common PTA balloon catheter (Active Comparator): use common PTA balloon catheter(trade name:Amphirion Deep) to treat stenosis or occlusion in below popliteal artery of control group
  Interventions: Procedure: common PTA balloon catheter

INTERVENTIONS:
Procedure: DEB catheter — DEB catheter (trade name: Litos/Tulip)
  Arms: DEB catheter
Procedure: common PTA balloon catheter — common PTA balloon catheter
  Arms: common PTA balloon catheter

SUMMARY:
The purpose of this study is to determine whether DEB is more effective than common PTA balloon using under in long-term vessel patency and inhibiting restenosis in the infrapopliteal artery.

DETAILED DESCRIPTION:
PTA is an established alternative to open surgical bypass for the treatment of infrainginual disease of critical limb ischemia.

DEBs are designed to promote arterial patency by reducing neointimal proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Patients with peripheral artery disease (PAD), with Rutherford classification between 4 and 6
* an occlusion or a minimum grade of stenosis Primary over 70% in the below popliteal artery
* The expected survival time is more than 1 year
* signed Patient informed consent form

Exclusion Criteria:

* Serum creatinine clearance rate less than 30ml/min in patients
* patients with acute thrombosis requiring lysis or thrombectomy
* patient with a lysis or an lower limb intervention as a therapy within the last 6 weeks
* patient requiring intervention in both lower limbs at the same time
* In-stent restenosis in the blow-knee popliteal artery
* target lesion can't be cross by the guide wire
* the stenosis rate of proximal outflow more than 30% with or without intervention
* the length of the stenosis or occlusion in proximal outflow(including the Iliac artery, the superficial femoral artery, the Popliteal artery) more than 150mm before intervention
* stenosis or occlusion of distal outflow for below-the-ankle artery.
* expected major amputations at the index limb before intervention
* known hypersensitivity to aspirin, heparin, clopidogrel,paclitaxel, contrast medium, etc.
* patients participating in another clinical trials with interfere with this trial in the same time
* pregnancy and lactating woman
* untreatable bleeding diatheses

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-05; Primary Completion 2018-11 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Primary Patency [Time Frame: 6 months] | 6 months
  Freedom from target vessel occlusion and clinically driven target lesion reintervention

SECONDARY OUTCOMES:
device success rate | during the operation(after using the DEB catheter)
  DEB catheter can reach the target lesions, expand as expected(not broken), and withdraw successfully.
technical success rates | during the operation(after using the DEB catheter)
  The blood supply of the target lesion recovered after treatment, and residual stenosis less than 50%
operation success rate | during the operation(after using the DEB catheter)
  both device succeed and technical succeed, and without clinical complication
if occured clinically driven TLR( target lesion revascularization) | 6 months, 12 months,18 months, 24 months
  Clinically driven TLR is defined as revascularization performed on a patient who returns with clinical symptoms such as: resting pain occur again, ulcer deterioration, new foot ulcers
target lesion late lumen loss 6 months | 6 months
  measure difference of the MLD(minimal lumen diameter) at 0 time and 6 months
Ulcer healing rate | 6 months, 12 months
  Healed or not, if not, improving,stagnant, worsening
Ulcer healing time | 6 months, 12 months, 18 months, 24 months
  Healed or not
Change from baseline ankle brachial index(ABI) at 6 months | 6 months
  measure ankle brachial index
  >1.3 Vascular wall calcification is severe
  0.9~1.1 Normal range
  0.5~0.8 Mild and moderate ischemia of lower limb arteries
  <0.5 severe ischemia
change from baseline Rutherford stage at 6 months | 6 months, 12 months,18 months, 24 months
  based the following definition of Rutherford stage, evaluate the stage of patient. Then compare the stage of patient just after procedure and 6 months after treatment
  Stage clinical symptom
  0 asymptomatic
  1. mild claudication
  2. moderate claudication
  3. severe claudication
  4. ischemic rest pain
  5. minor tissue loss
  6. ulceration or gangrene
limb salvage in surviving subjects | 30 days, 6 months, 12 months,18 months, 24 months
  No Amputation of target limb

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Chinese PLA General Hospital
Locations (11):
- China (11):
  - People's Liberation Army General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin

REFERENCES:
- [Derived] Jia X, Zhuang B, Wang F, Gu Y, Zhang J, Lu X, Dai X, Liu Z, Bi W, Liu C, Wang S, Liistro F, Guo W. Drug-Coated Balloon Angioplasty Compared With Uncoated Balloons in the Treatment of Infrapopliteal Artery Lesions (AcoArt II-BTK). J Endovasc Ther. 2021 Apr;28(2):215-221. doi: 10.1177/1526602820969681. Epub 2020 Oct 29. PMID 33118432